CLINICAL TRIAL: NCT07210970
Title: Study of The Prevalence of Latent Tuberculosis Infection Among Hemodialysis Patients Using Tuberculin Skin Test at Sohag University Hospital
Brief Title: Prevalence of Latent Tuberculosis Infection Among Hemodialysis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Ibrahim, Fatma Ahmed Ibrahim, Sohag University
Other Study IDs: Soh-Med--25-9-5MS
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Latent Tuberculosis Infection; End Stage Renal Disease (ESRD); Hemodialysis
MeSH Terms: conditions — Latent Tuberculosis; Kidney Failure, Chronic | interventions — Tuberculin Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodialysis Patients: Adult patients undergoing regular hemodialysis at Sohag University Hospital who will be screened for latent tuberculosis infection.
  Interventions: Diagnostic Test: Tuberculin Skin Test (TST)

INTERVENTIONS:
Diagnostic Test: Tuberculin Skin Test (TST) — Intradermal injection of 5 unit (0.1 mm) of purified protein derivative (PPD) with measurement of induration after 48-72 hours.

SUMMARY:
This observational cross-sectional study aims to determine the prevalence of latent tuberculosis infection (LTBI) among patients undergoing regular hemodialysis at Sohag University Hospital, using the tuberculin skin test (TST). Identifying the burden of LTBI in this high-risk population will help guide early detection and preventive strategies

DETAILED DESCRIPTION:
Patients receiving chronic hemodialysis are at increased risk of developing tuberculosis due to impaired immune function and frequent exposure to healthcare environments. Latent tuberculosis infection (LTBI) is particularly concerning in this population as it may progress to active disease, leading to increased morbidity and mortality. Early detection of LTBI among hemodialysis patients is essential to reduce this risk.

This cross-sectional study will be conducted at Sohag University Hospital. Two step tuberculin skin test (TST) will be administered to eligible adult patients undergoing regular hemodialysis, the first injection sitewill be examined between 48to 72 hours, and if negative, asecond booster injection will be given 1 to 2 weeks later. The prevalence of LTBI will be assessed by calculating the percentage of patients with a positive TST result (induration ≥10 mm ). Secondary analyses will examine associations between TST positivity and demographic or clinical variables, including age, sex, duration of dialysis, and comorbidities. The results are expected to contribute to local data on the burden of LTBI and to support preventive healthcare strategies in this vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Patients on regular hemodialysis Able and willing to provide informed consent

-

Exclusion Criteria:

* active TB patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing regular hemodialysis at Sohag University Hospital. The study will include patients aged 18 years and older who are clinically stable and able to undergo tuberculin skin testing
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of latent tuberculosis infection among hemodialysis patients. | Within 72 hours after TST administration.
  Percentage of patients with positive tuberculin skin test (defined as induration ≥10 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Fatma A Ibrahim, MSc, Principal Investigator — Faculty of Medicine, Sohag University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only aggregated results will be presented in the thesis and any related publications.